CLINICAL TRIAL: NCT04643522
Title: Does COVID-19 Worsen the Semen Parameters? Early Results of a Tertiary Health Center
Brief Title: Semen Parameters and COVID-19 in Infertile Men
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Erdem Koç, Medical Doctor, Ankara City Hospital Bilkent
Other Study IDs: E1-20-1237
Record Dates: First submitted 2020-11-24; First posted 2020-11-25 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Sperm Count, Low; Hormone Disturbance; Covid19
Keywords: COVID-19; Male infertility; Semen parameters; Sex-related hormone levels
MeSH Terms: conditions — Oligospermia; Endocrine System Diseases; COVID-19; Infertility, Male

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before COVID-19: The semen parameters and sex-related hormone levels of the patients which were performed before the diagnosis of COVID-19.
  Interventions: Other: Clinical assessment
- After COVID-19: The semen parameters and sex-related hormone levels of the patients which were performed after the diagnosis of COVID-19.
  Interventions: Other: Clinical assessment

INTERVENTIONS:
Other: Clinical assessment — Comparison of semen analysis results and sex-related hormone levels between the dependent groups which were defined as before COVID-19 and after COVID-19 (the data of the same patient group were compared as before and after the diagnosis of COVID-19).

SUMMARY:
Coronavirus Disease-19 (COVID-19) is a global pandemics which affects many organs and systems with a range of morbidities and high mortality rates. There are a number of studies revealed that COVID-19 may affect the testes and male genital tract which may in turn disrupt the gonadal functions.The current study aimed to evaluate the effect of COVID-19 on semen parameters and sex-related hormone levels.

DETAILED DESCRIPTION:
In this current study, the investigators aimed to elucidate the alteration in semen parameters of the infertile male patients who had been infected with SARS-CoV-2, through the comparison of the spermiogram results which were reported before and after the diagnosis of COVID-19. The investigators also aimed to evaluate the impact of COVID-19 on the sex-related hormone levels as follicle-stimulating hormone (FSH), luteinizing hormone (LH), and testosterone (T). The current study is conducted in Ankara City Hospital, the highest capacity tertiary health care center of the capital town of Turkey. The study included 21 patients who applied to Ankara City Hospital, Andrology Clinic for male infertility up to 05 October, 2020 and have had the semen analyses reported before and after the clinically confirmed diagnosis of COVID-19 through reverse transcriptase PCR. Besides the semen analyses, 8 of these 21 patients have also the had the reported levels of T, FSH and LH which were also analyzed.

ELIGIBILITY:
Inclusion Criteria:

Reproductive age Infertile men Clinically confirmed (with reverse transcriptase polymerase chain reaction-RT PCR) COVID-19 history Semen analyses performed before and after the diagnosis of COVID-19 (must be applicable for all patients) Sex-related hormone levels including FSH, LH, and T which were reported before and after the diagnosis of COVID-19 (was applicable for some of the patients)

Exclusion Criteria:

Azoospermia Semen analyses performed only before or after the diagnosis of COVID-19 Semen analysis performed in another hospital RT-PCR results which were reported in another hospital Chronical renal disease Chronical liver failure Patient age lower than 18 years old

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: The data of overall 25 patients who applied to our clinic for infertility evaluation and have had the semen analysis results reported before, and after the diagnosis of COVID-19 were reviewed. The 4 of the patients were found to have azoospermia. Due to the difficulty to compare the change at semen parameters in case of azoospermia as before and after results, these 4 patients were excluded. The study included 21 patients in final analyses. The results were presented through the two dependent group analyses, based on the patients' data collected before and after the diagnosis of COVID-19.
  The diagnosis of COVID-19 had been established according to the detection of SARS-CoV-2 in the sample taken from nasopharynx with a cotton swap, which was examined through the RT-PCR. None of the patients were at active phase of the COVID-19 at time of the semen sampling.The serum samples for hormone analyses were obtained on the same days with the semen samplings.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-10-10 (Actual)

PRIMARY OUTCOMES:
Semen analyses parameters including sperm motility (total, progressive, non-progressive and immotile | first 1 hour
  cell count percentage
Semen analyses parameters including sperm concentration | first 1 hour
  cell count per milliliters of semen sample.
Semen analyses parameters including sperm morphology | first 1 hour
  percentage of normal forms
Semen analyses parameters including semen volume | first 1 hour
  milliliters

SECONDARY OUTCOMES:
Sex-related hormone levels including testosterone | 20 minutes
  nanograms per deciliter
Sex-related hormone levels including follicle stimulating hormone and luteinizing hormone | 20 minutes
  Units per liter

CONTACTS AND LOCATIONS:
Overall Officials: Erdem Koç, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data belonging to participants will be available to any researcher or editorial reviewer board if needed.

REFERENCES:
- [Result] Holtmann N, Edimiris P, Andree M, Doehmen C, Baston-Buest D, Adams O, Kruessel JS, Bielfeld AP. Assessment of SARS-CoV-2 in human semen-a cohort study. Fertil Steril. 2020 Aug;114(2):233-238. doi: 10.1016/j.fertnstert.2020.05.028. Epub 2020 May 29. PMID 32650948
- [Result] Ma L, Xie W, Li D, Shi L, Ye G, Mao Y, Xiong Y, Sun H, Zheng F, Chen Z, Qin J, Lyu J, Zhang Y, Zhang M. Evaluation of sex-related hormones and semen characteristics in reproductive-aged male COVID-19 patients. J Med Virol. 2021 Jan;93(1):456-462. doi: 10.1002/jmv.26259. Epub 2020 Jul 19. PMID 32621617
- [Result] Achua JK, Chu KY, Ibrahim E, Khodamoradi K, Delma KS, Iakymenko OA, Kryvenko ON, Arora H, Ramasamy R. Histopathology and Ultrastructural Findings of Fatal COVID-19 Infections on Testis. World J Mens Health. 2021 Jan;39(1):65-74. doi: 10.5534/wjmh.200170. Epub 2020 Nov 3. PMID 33151050
- [Result] Yang M, Chen S, Huang B, Zhong JM, Su H, Chen YJ, Cao Q, Ma L, He J, Li XF, Li X, Zhou JJ, Fan J, Luo DJ, Chang XN, Arkun K, Zhou M, Nie X. Pathological Findings in the Testes of COVID-19 Patients: Clinical Implications. Eur Urol Focus. 2020 Sep 15;6(5):1124-1129. doi: 10.1016/j.euf.2020.05.009. Epub 2020 May 31. PMID 32563676